CLINICAL TRIAL: NCT04306172
Title: External Validation of EPIC's Readmission Risk Model, the LACE+ Index and SQLape as Predictors of Unplanned Hospital Readmissions: A Monocentric, Retrospective, Diagnostic Cohort Study in Switzerland
Brief Title: Validation of EPIC's Readmission Risk Model, the LACE+ Index and SQLape as Predictors of Unplanned Hospital Readmissions
Status: Completed | Type: Observational
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Universität Luzern (Other)
Responsible Party: Principal Investigator, Aljoscha Hwang, Research Project Manager & Advanced Analytics Analyst, Luzerner Kantonsspital
Other Study IDs: LUKS_RRM_2019
Record Dates: First submitted 2020-03-06; First posted 2020-03-12 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Hospital Readmission
Keywords: Prediction model; hospital readmission; external validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Readmitted inpatients/Cases: Outcome 1: Patients who were readmitted within 18 days of index hospitalization discharge date to the same hospital, with a diagnosis leading to the same Major Diagnostic Group as the index stay (definition according to Swiss Diagnosis Related Groups system, case merger)
  Outcome 2: Patients with an unplanned readmission within 30 days of index hospitalization discharge date to the same hospital. An unplanned readmission was defined as a readmission through the emergency department.
  Interventions: Other: An US Readmission Risk Prediction Model; Other: LACE+ score; Other: SQLAPE model
- Non-Readmitted inpatients/Controls: Outcome 1 & 2: Patients who were not readmitted within 30 days of index hospitalization discharge date.
  Interventions: Other: An US Readmission Risk Prediction Model; Other: LACE+ score; Other: SQLAPE model

INTERVENTIONS:
Other: An US Readmission Risk Prediction Model — Logistic regression model that predicts the risk of all-cause unplanned readmissions developed by the privately held healthcare software company EPIC.
Other: LACE+ score — The LACE+ score is a point score that can be used to predict the risk of post-discharge death or urgent readmission. It was developed based on administrative data in Ontario, Canada.
Other: SQLAPE model — The readmission risk model (Striving for Quality Level and analyzing of patient expenditures), is a computerized validated algorithm and was developed in 2002 to identify potentially avoidable readmissions.

SUMMARY:
The primary objective of this study is to externally validate the EPIC's Readmission Risk model and to compare it with the LACE+ index and the SQLape Readmission model.

As secondary objective, the EPIC's Readmission Risk model will be adjusted based on the validation sample, and finally, it´s performance will be compared with machine learning algorithms.

DETAILED DESCRIPTION:
Introduction: Readmissions after an acute care hospitalization are relatively common, costly to the health care system and are associated with significant burden for patients. As one way to reduce costs and simultaneously improve quality of care, hospital readmissions receive increasing interest from policy makers. It is only relatively recently that strategies were developed with the specific aim of reducing unplanned readmissions by applying prediction models. EPIC's Readmission Risk model, developed in 2015 for the U.S. acute care hospital setting, promises superior calibration and discriminatory abilities. However, its routine application in the Swiss hospital setting requires external validation first. Therefore, the primary objective of this study is to externally validate the EPIC's Readmission Risk model and to compare it with the LACE+ index (Length of stay, Acuity, Comorbidities, Emergency Room visits index) and the SQLape (Striving for Quality Level and analysing of patient expenditures) Readmission model.

Methods: For this reason, a monocentric, retrospective, diagnostic cohort study will be conducted. The study will include all inpatients, who were hospitalized between the 1st January 2018 and the 31st of January 2019 in the Lucerne Cantonal hospital in Switzerland. Cases will be inpatients that experienced an unplanned (all-cause) readmission within 18 or 30 days after the index discharge. The control group will consist of individuals who had no unscheduled readmission.

For external validation, discrimination of the scores under investigation will be assessed by calculating the area under the receiver operating characteristics curves (AUC). For calibration, the Hosmer-Lemeshow goodness-of-fit test will be graphically illustrated by plotting the predicted outcomes by decile against the observations. Other performance measures to be estimated will include the Brier Score, Net Reclassification Improvement (NRI) and the Net Benefit (NB).

All patient data will be retrieved from clinical data warehouses.

ELIGIBILITY:
Inclusion Criteria:

- All inpatients, aged one year or older (max. 100 years), who were hospitalized either between the 1st of January 2018 and the 31st of December 2018, or between the 23rd of September and the 31st of December 2019 will be included.

Exclusion criteria:

* admission/transfer from another psychiatric, rehabilitative or acute care ward from the same institution,
* discharge destination other than the patient's home or
* transfer to another acute care hospital, both being considered as treatment continuation;
* foreign residence,
* deceased before discharge,
* discharged on admission day,
* refusal of general consent, and
* unknown patient residence or discharge destination.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients from an acute care hospital in Central-Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 23116 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Discrimination at 18 days | 18 days after index discharge date
  For discrimination of the scores under investigation, the area under the receiver operating characteristics curves (AUC) will be calculated.
Discrimination at 30 days | 30 days after index discharge date
  For discrimination of the scores under investigation, the area under the receiver operating characteristics curves (AUC) will be calculated.
Calibration at 18 days | 18 days after index discharge date
  For calibration, the Hosmer-Lemeshow goodness-of-fit test will be graphically illustrated by plotting the predicted outcomes by decile against the observations.
Calibration at 30 days | 30 days after index discharge date
  For calibration, the Hosmer-Lemeshow goodness-of-fit test will be graphically illustrated by plotting the predicted outcomes by decile against the observations.
Overall Performance at 18 days | 18 days after index discharge date
  Brier Score (The Brier score is a quadratic scoring rule, where the squared difference between actual binary outcomes Y and predictions p are calculated. The Brier score can range from 0 for a perfect model to 0.25 for a non-informative model with a 50% incidence of the outcome.)
Overall Performance at 30 days | 30 days after index discharge date
  Brier Score (The Brier score is a quadratic scoring rule, where the squared difference between actual binary outcomes Y and predictions p are calculated. The Brier score can range from 0 for a perfect model to 0.25 for a non-informative model with a 50% incidence of the outcome.)
Clinical usefulness (NRI) at 18 days | 18 days after index discharge date
  Net Reclassification Improvement (NRI): In the calculation of the NRI, the improvement in sensitivity and the improvement in specificity are summed. The NRI ranges from 0 for no improvement and 1 for perfect improvement.
Clinical usefulness (NRI) at 30 days | 30 days after index discharge date
  Net Reclassification Improvement (NRI): In the calculation of the NRI, the improvement in sensitivity and the improvement in specificity are summed. The NRI ranges from 0 for no improvement and 1 for perfect improvement.
Clinical usefulness (NB) at 18 days | 18 days after index discharge date
  Net Benefit (NB): NB = (TP - w FP) / N, where TP is the number of true positive decisions, FP the number of false positive decisions, N is the total number of patients and w is a weight equal to the odds of the cut-off (pt/(1-pt), or the ratio of harm to benefit
Clinical usefulness (NB) at 30 days | 30 days after index discharge date
  Net Benefit (NB): NB = (TP - w FP) / N, where TP is the number of true positive decisions, FP the number of false positive decisions, N is the total number of patients and w is a weight equal to the odds of the cut-off (pt/(1-pt), or the ratio of harm to benefit

CONTACTS AND LOCATIONS:
Overall Officials: Aljoscha B. Hwang, Principal Investigator — University Lucerne (Switzerland); Stefan Boes, Principal Investigator — University Lucerne (Switzerland)
Locations (1):
- Cantonal Hospital of Lucerne, Lucerne, Canton Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Walraven C, Wong J, Forster AJ. LACE+ index: extension of a validated index to predict early death or urgent readmission after hospital discharge using administrative data. Open Med. 2012 Jul 19;6(3):e80-90. Print 2012. PMID 23696773
- [Background] Halfon P, Eggli Y, Pretre-Rohrbach I, Meylan D, Marazzi A, Burnand B. Validation of the potentially avoidable hospital readmission rate as a routine indicator of the quality of hospital care. Med Care. 2006 Nov;44(11):972-81. doi: 10.1097/01.mlr.0000228002.43688.c2. PMID 17063128

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT04306172/Prot_SAP_000.pdf